CLINICAL TRIAL: NCT06561451
Title: A Randomized Control Trial to Compare the Live Birth Rate Between Intracytoplasmic Sperm Injection and Artificial Oocyte Activation and Intracytoplasmic Sperm Injection Alone in Patients With Severe Teratospermia
Brief Title: Live Birth Rate Between ICSI and AOA and ICSI Alone in Patients With Severe Teratospermia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ShangHai Ji Ai Genetics & IVF Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JIAI 2024-08
Record Dates: First submitted 2024-08-17; First posted 2024-08-20 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Male Infertility; Teratospermia
MeSH Terms: conditions — Infertility, Male; Teratozoospermia | interventions — Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICSI+AOA group (Experimental): ICSI+AOA group: a single sperm will be injected within 4 hours after the follicular aspiration. All injected oocytes will be incubated in the calcium ionophore A23187 activation solution (C9275-1MG, Sigma, USA) for 10 min, and cultured in the cleavage medium (Cleavage Medium , Cook, United States) under standard conditions.
  Interventions: Procedure: intracytoplasmic sperm injection and artificial oocyte activation
- ICSI group (Active Comparator): a single sperm will be injected within 4 hours after the follicular aspiration.
  Interventions: Procedure: intracytoplasmic sperm injection

INTERVENTIONS:
Procedure: intracytoplasmic sperm injection and artificial oocyte activation — A single sperm will be injected within 4 hours after the follicular aspiration. All injected oocytes will be incubated in the calcium ionophore A23187 activation solution (C9275-1MG, Sigma, USA) for 10 min, and cultured in the cleavage medium (Cleavage Medium , Cook, United States) under standard conditions.
  Arms: ICSI+AOA group
Procedure: intracytoplasmic sperm injection — A single sperm will be injected within 4 hours after the follicular aspiration.
  Arms: ICSI group

SUMMARY:
The goal of this clinical trial is to compare the live birth rate between intracytoplasmic sperm injection (ICSI) and artificial oocyte activation (AOA) vs intracytoplasmic sperm injection alone in patients with teratospermia. The hypothesis is the live birth rate following ICSI and AOA is significantly higher than that by ICSI alone in patients with teratospermia. This is a randomized controlled trial. Participants will be randomly assigned into one of the two groups:

ICSI+AOA group: a single sperm will be injected within 4 hours after the follicular aspiration. All injected oocytes will be incubated in the calcium ionophore A23187 activation solution (C9275-1MG, Sigma, USA) for 10 min, and cultured in the cleavage medium (Cleavage Medium , Cook, United States) under standard conditions.

ICSI alone group: a single sperm will be injected within 4 hours after the follicular aspiration.

ELIGIBILITY:
Inclusion Criteria:

1. Age of women 20-37 years at the time of ovarian stimulation for ICSI
2. At least three matured oocytes Severe teratozoospermia: defined as abnormal sperm morphology ranging between 99-100%, including globozoospermia and tapered-head.

Exclusion Criteria:

1. Presence of hydrosalpinx which is not surgically treated
2. Undergoing preimplantation genetic testing
3. Recurrent pregnancy loss (defined as two or more previous spontaneous pregnancy losses)
4. Known uterine abnormality (e.g., uterine congenital malformation; untreated uterine septum, adenomyosis, or submucous myoma; endometrial polyps; or intrauterine adhesions)
5. Abnormal parental karyotyping, or Medical conditions that assisted reproductive technology or pregnancy is contraindicated

Ages: 20 Years to 37 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 208 (Estimated)
Dates: Start 2024-08-30 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Live birth | 1 year after embryo transfer
  Delivery ≥22 weeks of gestation with heartbeat and breath.

SECONDARY OUTCOMES:
Fertilization rate | 1 day after oocyte retrieval
  Fertilized oocytes with two pronuclei per MII oocyte injected
High-quality embryos on Day 3 | 3 days after oocyte retrieval
  Seven or eight blastomeres of equal-size and <20% fragmentation by volume
hCG positivity | 14 days after embryo transfer
  Serum hCG level ≥10mIU/mL
Number and grading of embryos/blastocysts | 6 days after oocyte retrieval
  Number and grading of embryos/blastocysts suitable for freezing and transfer
Clinical pregnancy | 6 weeks of gestation
  the presence of an intrauterine gestational sac on transvaginal ultrasound at 6 gestational weeks.
Ongoing pregnancy | 12 weeks of gestation
  a viable pregnancy beyond 12 weeks of gestation
Multiple pregnancy | 6 weeks of gestation
  presence of more than one intrauterine sac at 6 weeks of gestation
Cumulative live birth rate (within 6 months after randomization) | 1.5 years after the randomization
  Any live birth arising from embryo transfer within 6 months after randomization
Miscarriage rate | 22 weeks of pregnancy
  A clinically recognized pregnancy loss before 22 weeks of pregnancy. The denominator is the clinical pregnancy.
Birth weights of the newborns | 1 year after embryo transfer
  Birth weights of the newborns

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoxi Sun, PhD, Study Director — Shanghai JiAi Genetics & IVF Institute
Locations (1):
- ShangHai JIAI Genetics &I VF Institute, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Data from the trial will be shared according to the International Committee of Medical Journal Editors guidelines. Individual participant data that underlie the results after deidentification (text, tables, figures and appendices) and the study protocol will be shared. On request, data can be shared with parties presenting relevant aims for the use of data. Data will be available from 3 months to 5 years following article publication.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available from 3 months to 5 years following article publication
Access Criteria: On request, data can be shared with parties presenting relevant aims for the use of data. Please contact the researcher through email: lihe198900@163.com.

REFERENCES:
- [Background] Palermo G, Joris H, Devroey P, Van Steirteghem AC. Pregnancies after intracytoplasmic injection of single spermatozoon into an oocyte. Lancet. 1992 Jul 4;340(8810):17-8. doi: 10.1016/0140-6736(92)92425-f. PMID 1351601
- [Background] Yeste M, Jones C, Amdani SN, Patel S, Coward K. Oocyte activation deficiency: a role for an oocyte contribution? Hum Reprod Update. 2016 Jan-Feb;22(1):23-47. doi: 10.1093/humupd/dmv040. Epub 2015 Sep 7. PMID 26346057
- [Background] Van Steirteghem AC, Nagy Z, Joris H, Liu J, Staessen C, Smitz J, Wisanto A, Devroey P. High fertilization and implantation rates after intracytoplasmic sperm injection. Hum Reprod. 1993 Jul;8(7):1061-6. doi: 10.1093/oxfordjournals.humrep.a138192. PMID 8408487
- [Background] De Vos A, Van De Velde H, Joris H, Verheyen G, Devroey P, Van Steirteghem A. Influence of individual sperm morphology on fertilization, embryo morphology, and pregnancy outcome of intracytoplasmic sperm injection. Fertil Steril. 2003 Jan;79(1):42-8. doi: 10.1016/s0015-0282(02)04571-5. PMID 12524062
- [Background] Lu YH, Gao HJ, Li BJ, Zheng YM, Ye YH, Qian YL, Xu CM, Huang HF, Jin F. Different sperm sources and parameters can influence intracytoplasmic sperm injection outcomes before embryo implantation. J Zhejiang Univ Sci B. 2012 Jan;13(1):1-10. doi: 10.1631/jzus.B1100216. PMID 22205614
- [Background] Greco E, Scarselli F, Fabozzi G, Colasante A, Zavaglia D, Alviggi E, Litwicka K, Varricchio MT, Minasi MG, Tesarik J. Sperm vacuoles negatively affect outcomes in intracytoplasmic morphologically selected sperm injection in terms of pregnancy, implantation, and live-birth rates. Fertil Steril. 2013 Aug;100(2):379-85. doi: 10.1016/j.fertnstert.2013.04.033. Epub 2013 May 23. PMID 23706334
- [Background] Vanden Meerschaut F, Nikiforaki D, Heindryckx B, De Sutter P. Assisted oocyte activation following ICSI fertilization failure. Reprod Biomed Online. 2014 May;28(5):560-71. doi: 10.1016/j.rbmo.2014.01.008. Epub 2014 Jan 31. PMID 24656559
- [Background] Vanden Meerschaut F, Nikiforaki D, De Gheselle S, Dullaerts V, Van den Abbeel E, Gerris J, Heindryckx B, De Sutter P. Assisted oocyte activation is not beneficial for all patients with a suspected oocyte-related activation deficiency. Hum Reprod. 2012 Jul;27(7):1977-84. doi: 10.1093/humrep/des097. Epub 2012 Apr 4. PMID 22493027